CLINICAL TRIAL: NCT01984112
Title: Proximal Humerus Fractures: Randomized Study Between Intramedullary Locking Nails and Locking Plates for Neer 2 and 3 Parts Displaced Fractures
Brief Title: Proximal Humerus Fractures: Randomized Study Between Locking Nails and Locking Plates for Neer 2 and 3 Parts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mauro Gracitelli, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0232/11
Record Dates: First submitted 2013-10-28; First posted 2013-11-14 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Humerus; Proximal Humeral Fracture; Fractures, Bone; Humeral Fractures; Wounds and Injuries; Arm Injuries
Keywords: Humerus; fracture; nail; plate; tuberosity
MeSH Terms: conditions — Shoulder Fractures; Fractures, Bone; Humeral Fractures; Wounds and Injuries; Arm Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramedullary Locked Nail (Experimental)
  Interventions: Device: Intramedullary locked nail
- Locked Plate (Active Comparator)
  Interventions: Device: Locked plate

INTERVENTIONS:
Device: Locked plate — Osteosynthesis with philos plate, through deltopectoral approach and rotator cuff augmentation with inabsorbable poliester suture
  Other Names: Philos plaste, Synthes, Switzerland
  Arms: Locked Plate
Device: Intramedullary locked nail — Intramedullary locked nail performed by antero-lateral transdeltoid minimally invasive approach and rotator cuff augmentation with inabsorbable poliester suture
  Other Names: Centronail, Proximal Humeral Nail, Orthofix, Italy
  Arms: Intramedullary Locked Nail

SUMMARY:
The hypothesis of this study is to determine whether the technique of intramedullary locking nail presents clinical results comparable to the technique of locking plates, based on the Constant Score.

ELIGIBILITY:
Inclusion Criteria:

* Fracture with less than 21 days;
* Fractures of the proximal humerus classified as 2 or 3 parts of Neer, with involvement of the humeral head and one of the tuberosities;
* Fracture with unacceptable deviation for the non-surgical treatment, according to the criteria of Neer Neer: fractures with deviation greater than 45 ° or 1 cm for the fragment of the humeral head and fractures with a deviation of the tuberosity greater than 0.5 cm;
* Closed fractures;

Exclusion Criteria:

* Characteristics of the fracture:

  * fracture between the greater tubercle and the smaller, independent of the deviation;
  * Isolated fracture of the greater or lesser tuberosity
  * 4-part fractures of Neer;
  * Fracture involving the articular surface of the humeral head;
  * Fracture-dislocation of the proximal humerus
* Other criteria:

  * Neurological injuries in the affected limb;
  * previous surgery on the affected shoulder;
  * associated fractures in the affected limb;
  * pathologic fractures;
  * lesions of the rotator cuff tendons previously diagnosed;
  * Psychiatric illnesses or inability to understand preoperative questionnaires;
  * Active infection or previous infection on the shoulder;

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Shoulder function, pain, strength and range of motion, measured by Constant-Murley Score | 12 months
  Absolute Constant-Murley Score, that measures:
  Shoulder function, pain, strength and range of motion 0-100 points score 12 months as the final outcome

SECONDARY OUTCOMES:
Superior limb function, measured by DASH score | 12 months
  Disability of Arm-Shoulder-Hand score
Shoulder function, pain, strength, range of motion and satisfaction with treatment, measured by UCLA score | 12 months
  Shoulder function, pain, strength, range of motion and satisfaction with treatment, measured by University of California Los Angeles score.
  0-35 points score
Shoulder function, pain, strength and range of motion compared with non-injuried shoulder, measured by Individual Relative Constant-Murley Score | 12 months
  Individual Relative Constant-Murley Score, compared to non-injured shoulder.
  Fialka C, Oberleitner G, Stampfl P, Brannath W, Hexel M, Vécsei V. Modification of the Constant-Murley shoulder score-introduction of the individual relative Constant score Individual shoulder assessment. Injury. 2005 Oct;36(10):1159-65.
Number of patients with complications | 12 months
  Overall complications and need for additional surgery, categorized as:
  Not related to implant
  Clinical
  * Death in the intraoperative or postoperative period;
  * Clinical complications related to surgery .
  Orthopedic
  * Infection
  * Osteonecrosis ;
  * Nonunion ;
  * Stiffness
  * Reflex sympathetic dystrophy ;
  * Heterotopic ossification ;
  * Refracture ;
  * Neurological injury .
  * Insufficient reduction;
  * Loss of reduction of the humeral head;
  * Loss of reduction of tubercule: deviation greater than 5 mm between the immediate postoperative radiographs and 12 months;
  Related to the implant
  * Primary articular protrusion of screws;
  * Loosening of the implant ;
  * Breaking of the implant ;
  * Cutout: loss reduction head with proximal screw pullout ;
  * secondary articular protrusion screws;
  * Malunion
  * Injury to the rotator cuff tendons is observed in postoperative ultrasonography;

OTHER OUTCOMES:
Post-operative integrity of the rotator cuff, evaluated by ultrasonography | 6 months
  Post-operative integrity of the rotator cuff, evaluated by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Mauro EC Gracitelli, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196